CLINICAL TRIAL: NCT03064646
Title: ORGAN PRESERVATION AFTER NEOADJUVANT TREATMENT FOR LOCALLY ADVANCED RECTAL CANCER
Brief Title: Organ Preservation in Locally Advanced Rectal Cancer
Acronym: PRONAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Javier Gallego Plazas, PhD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRONAR V1.0: 19DEC2016
Record Dates: First submitted 2017-02-16; First posted 2017-02-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: LOCALLY ADVANCED RECTAL CANCER
Keywords: ORGAN PRESERVATION; WATCH AND WAIT; TRANSANAL ENDOSCOPIC MICROSURGERY
MeSH Terms: interventions — Organ Preservation; Transanal Endoscopic Microsurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organ Preservation (Experimental): The experimental strategy is the omission of radical surgery if complete or almost complete response after neoadjuvant treatment for locally advanced rectal cancer
  Interventions: Other: Organ Preservation

INTERVENTIONS:
Other: Organ Preservation — Patients with a complete response or a almost complete response after neoadjuvant treatment will be offered an organ preservation strategy
  Other Names: Transanal Endoscopic Microsurgery; Watch and Wait

SUMMARY:
PRONAR trial aims to assess if treatment with organ preservation in stage II and III rectal cancer after a complete or almost complete response to neoadjuvant treatment is feasible and safe in our environment.

The main objective of this project is to implement the organ preservation strategy in the treatment of rectal cancer in our environment within a clinical study that allows the analysis of its results in terms of survival.

The secondary objective is to assess local relapse, distant relapse and quality of life.

DETAILED DESCRIPTION:
After pathology confirmed rectal cancer patients with stage II and III (MRI, CT and endoscopy) will be identified in the first visit to Medical Oncology Department. Patients will receive the most appropriate neoadjuvant treatment according to clinical guidelines.

Response to neoadjuvant treatment will be assessed by MRI. Those patients with a complete response in MRI, confirmed by endoscopy, will be offered a "watch and wait" strategy. Patients with a complete response in MRI, with an almost complete response in endoscopy, will be offered transanal endoscopic microsurgery. All patients with complete or near complete response will sign an informed consent before study entry.

Radical surgery will be performed in patients without complete or almost complete response criteria after neoadjuvant treatment.

Patients in organ preserving strategy will be subjected to a more intensive follow up schedule, including MRI and endoscopy, compared to patients with radical surgery.

As the complete histopathologic response rate after neoadjuvant treatment in locally advanced rectal cancer is approximately 15-20%, considering that approximately 40 patients with locally advanced rectal cancer are diagnosed annually in our setting, approximately 6-8 patients per year could be potentially recruited for this project, until reaching an initial sample of 30 patients for evaluation.

The following results will be analyzed:

* Percentage of complete and almost complete responses.
* Percentage of watch and wait and transanal endoscopic microsurgery.
* Disease free survival.
* Overall survival.
* Local relapse rate.
* Distant relapse rate.
* Treatment and outcomes of relapses.
* Colostomy free survival.
* Quality of life.

All data will be obtained from patient's medical records

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed histopathological diagnosis of rectal adenocarcinoma.
* Patients treated with neoadjuvant chemoradiotherapy or neoadjuvant radiotherapy associated or not with induction chemotherapy.
* Patients with evidence of complete or near complete response criteria after completion of neoadjuvant treatment (approximately 8 weeks later). Response criteria should be based on digital rectal examination, flexible rectoscopy and MRI.

Exclusion Criteria:

* Evidence of distant metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of organ preservative strategies after neoadjuvant treatment in locally advanced rectal cancer | 5 years
  Patients with a complete or almost complete response after a neoadjuvant treatment will be offered an organ preservation strategy

SECONDARY OUTCOMES:
Local relapse rate | 2 years and 5 years
  Occurrence of local relapse in patients with an organ preservation strategy
Distant relapse rate | 2 years and 5 years
  Occurrence of distant relapse in patients with an organ preservation strategy
Quality of Life in oncological patients | 3 months; 1 year and annually until 5 years
  Assess QLQ-C30 in patients with an organ preservation strategy
Quality of Life in patient with rectal cancer | 3 months, 1 year and annually until 5 years
  Assess QLQ-CR38 in patients with an organ preservation strategy

OTHER OUTCOMES:
Percentage of complete and almost complete responses | 8 weeks after neoadjuvant treatment
  Occurrence of complete and almost complete responses assessed by MRI and confirmed by endoscopy after neoadjuvant treatment
Disease free survival | 2 years and 5 years
  Time without recidive
Overall Survival | 2 years and 5 years
  Survival time from surgery
Treatment of relapses | 2 years and 5 years
  Treatment administered in case of relapse
Outcome of relapses | 2 years and 5 years
  Survival after a relapse
Colostomy free survival | 2 years and 5 years
  Time without colostomy

CONTACTS AND LOCATIONS:
Overall Officials: Javier Gallego, PhD, Principal Investigator — Hospital General Universitario de Elche; Javier Gallego, PhD, Study Director — Hospital General Universitario de Elche
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
It is planned to share global data analysis